CLINICAL TRIAL: NCT04896099
Title: Prospective, Observational Study Evaluating the Feasibility of a Systematic and Standardized Assessment of Supportive Care Needs in Patients With Advanced Solid Cancer at the Inclusion in a Therapeutic Trial at the Institut Curie
Brief Title: Feasibility of Supportive Care Needs in Patients With Advanced Solid Cancer in a Therapeutic Trial
Acronym: ES4-UIC
Status: Completed | Type: Observational
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Other Study IDs: IC 2020-18
Record Dates: First submitted 2021-05-06; First posted 2021-05-21 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Supportive Care; Metastatic Cancer; Clinical Trial
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to assess the supportive care needs of patients enrolled in a therapeutic trial for metastatic cancer.

DETAILED DESCRIPTION:
All patients included in a therapeutic trial will be offered an analysis of their supportive care needs from the following options:

* dietetics
* psychological
* pain management
* Palliative medicine consultation or day hospital
* onco-geriatrics
* social assistance
* Physiotherapist care If an intervention(s) is selected, it will be offered in addition to the patient's participation in the therapeutic trial.

ELIGIBILITY:
Inclusion Criteria:

* metastatic cancer
* patient included in a clinical trial

Exclusion Criteria:

- patient deprived of his freedom

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all comers for a clinical trial
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
EORTC Core Quality of Life Questionnaire (EORTC QLQ-C30) | 3 months
  Descritive results with validated questionnaire for the assessment of Quality of life in patient with cancer. 30 Questions
National Comprehensive Cancer Network (NCCN) Distress thermometer | 3 months
  Descritive results with validated questionnaire for distress assessment (scale from 0 to 10 and list of problems to be ticked by the patient
Questionnaire G8 oncodage | 3 months
  Descritive results with validated questionnaire for the identification of geriatric frailties in 70 year old cancer patients. Score on 17 points: > 14 = standard care, <14 = specialized geriatric evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Pauline du Rusquec, MD, Principal Investigator — Institut Curie
Locations (1):
- Institut Curie, Paris, France